CLINICAL TRIAL: NCT02684877
Title: Fatigue in Intensive Care Survivors One Year After Discharge
Brief Title: Fatigue One Year After ICU Discharge
Status: Completed | Type: Observational
Sponsor: Università degli Studi di Ferrara (Other)
Responsible Party: Principal Investigator, Savino Spadaro, Physician, Università degli Studi di Ferrara
Other Study IDs: fatigue
Record Dates: First submitted 2016-02-13; First posted 2016-02-18 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-04

CONDITIONS: Fatigue
Keywords: Fatigue; Quality of life; Critically ill patients
MeSH Terms: conditions — Fatigue | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Intensive care survivors: Observational study
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire

SUMMARY:
The investigators contacted consecutive adult patients admitted to intensive care unit (ICU) and mechanically ventilated for at least 72 hours to invite them to an interview at hospital. The investigators administered Mini Mental Status Examination, Functional Assessment of Chronic Illness Therapy scale for Fatigue (Facit- F) and Short form 36 questionnaires to the consenting patients.

DETAILED DESCRIPTION:
Fatigue is one of the most commonly symptoms reported by patients. There are many causes of pathological fatigue including mental and physical, both neurological (central and peripheral) and non-neurological diseases. Among the last ones, cancer, infections and drugs are factors associated with fatigue, although the mechanism of how non-neurological diseases cause fatigue is not clear. Evidence exists to suggest that patients who have been critically ill continue to face a multitude of physical, psychological and social difficulties in the long term after discharge. As far as fatigue is concerned, greater than 50% of Intensive Care Unit survivors overall reported lowered energy levels and fatigue in the first year after discharge.

ELIGIBILITY:
Inclusion Criteria:

* aged > 18 years
* able to co-operate at the time of ICU discharge
* requiring mechanical ventilation for at least 72 hours
* residents less than 30 km from the hospital

Exclusion Criteria:

* preexisting cognitive deficits
* pre-existing psychotic illness
* admitted for anoxic brain injury
* residents more than 30 km from the hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intensive care one-year survivors
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2015-01; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Functional Assessment Chronic Illness Therapy-Fatigue (FACIT-F) | 12 months

SECONDARY OUTCOMES:
Short form 36 questionnaire | 12 months

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Finsterer J, Mahjoub SZ. Fatigue in healthy and diseased individuals. Am J Hosp Palliat Care. 2014 Aug;31(5):562-75. doi: 10.1177/1049909113494748. Epub 2013 Jul 26. PMID 23892338
- [Background] Apolone G, Mosconi P. The Italian SF-36 Health Survey: translation, validation and norming. J Clin Epidemiol. 1998 Nov;51(11):1025-36. doi: 10.1016/s0895-4356(98)00094-8. PMID 9817120
- [Background] Egerton T, Riphagen II, Nygard AJ, Thingstad P, Helbostad JL. Systematic content evaluation and review of measurement properties of questionnaires for measuring self-reported fatigue among older people. Qual Life Res. 2015 Sep;24(9):2239-55. doi: 10.1007/s11136-015-0963-1. Epub 2015 Mar 17. PMID 25778536
- [Derived] Spadaro S, Capuzzo M, Valpiani G, Bertacchini S, Ragazzi R, Dalla Corte F, Terranova S, Marangoni E, Volta CA. Fatigue in intensive care survivors one year after discharge. Health Qual Life Outcomes. 2016 Oct 18;14(1):148. doi: 10.1186/s12955-016-0554-z. PMID 27756403